CLINICAL TRIAL: NCT04002505
Title: Shared Decision Making for Patients With Minor Head Injury: The "Concussion or Brain Bleed" Trial
Brief Title: The "Concussion or Brain Bleed" Trial
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Neha P. Raukar, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-000224
Record Dates: First submitted 2019-06-27; First posted 2019-06-28 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Head Injury
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Head Injury Subject (Experimental): Subjects that present to the Emergency Department with a blunt head injury within the past 24 hours, determined to be low risk by the Canadian CT Head Rules (CCHR), and are being considered for a head CT by the treating provider will use the shared decision making tool Concussion and Brain Bleed app (CBC) with their clinician
  Interventions: Other: Concussion and Brain Bleed App (CBB)

INTERVENTIONS:
Other: Concussion and Brain Bleed App (CBB) — Tablet based decision aid that encourages shared decision making with the goal of educating patients to reduce unnecessary CT scans

SUMMARY:
Researchers are trying to understand the effect of educating patients and encouraging shared decision making on rates of CT scanning in head injured patients by using an already developed app and observing the effect on the health care provider.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Present to the Emergency Department with a blunt head injury within the past 24 hours
* Determined to be low risk by the Canadian CT Head Rules (CCHR), and are being considered for a head CT by the treating provider.

Exclusion Criteria:

* Patients who are pregnant
* Non-English speaking
* In police custody
* Undergoing psychiatric evaluation
* Found to have drug or alcohol intoxication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2019-06-27 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Rate of CT Scans | 6 months
  Number of CT scans performed when using the Concussion and Brain Bleed app

CONTACTS AND LOCATIONS:
Overall Officials: Neha Raukar, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials (open in google chrome) — https://www.mayo.edu/research/clinical-trials